CLINICAL TRIAL: NCT02031679
Title: A Phase IIa, Randomized, Placebo-controlled, Double-blind Study to Assess the Efficacy and Safety of the CRTh2 Antagonist AZD1981 in Patients With Chronic Idiopathic Urticaria (CIU) Who Are Refractory to H1 Antihistamines
Brief Title: Efficacy and Safety of Chemoattractant Receptor-homologous Molecule Expressed on T Helper Type 2 (CRTh2) Antagonist AZD1981 in Chronic Idiopathic Urticaria (CIU) Antihistamines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00089252
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Chronic Idiopathic Urticaria
Keywords: Chronic Idiopathic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — AZD1981

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD1981 (Experimental): AZD1981 for oral administration will be available in tablet form. AZD1981 tablets will be provided in 10 mg strengths.
  The drug will be self-administered by the subject. Subjects will take 4 tablets in the morning, 4 tablets in the afternoon, and 4 tablets in the evening.
  The tablets should be swallowed whole with a glass of water.
  Interventions: Drug: AZD1981
- Placebo (Placebo Comparator): The placebo will be available in tablet form. The placebo contains the same ingredients as the AZD1981 with the exception of the active compound.
  The placebo will be self-administered by the subject. Subjects will take 4 tablets in the morning, 4 tablets in the afternoon, and 4 tablets in the evening.
  The tablets should be swallowed whole with a glass of water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1981 — AZD1981 is an oral, potent, selective, reversible antagonist of CRTh2 (Chemoattractant Receptor Homologous Molecule expressed on Th2 cells).
  Other Names: Oral CRTh2 antagonist
  Arms: AZD1981
Drug: Placebo — Sugar pill manufactured to mimic AZD1981 10 mg tablet
  Arms: Placebo

SUMMARY:
The investigators are recruiting for a chronic hives study. This research is being done to test whether an investigational drug called AstraZeneca drug (AZD)1981 may be helpful for treating people with Chronic Idiopathic Urticaria who continue to have symptoms despite taking antihistamines. The word "investigational" means that AZD1981 is not approved for marketing by the Food and Drug Administration (FDA). The FDA is allowing the use of AZD1981 in this study.

People with chronic hives lasting for at least 6 months and without a known cause may join. The study involves 6 visits over 8 weeks. Approximately 48 participants expected to take part in this study at the Johns Hopkins Asthma and Allergy Clinic. All participants will be treated with the study medication and/or placebo for 8 weeks.

The results of this trial may have a benefit others with Chronic Idiopathic Urticaria who don't respond well to antihistamines by generating experience and data to support the design of a larger, multicenter trial investigating the efficacy of AZD1981 in treating antihistamine refractory CIU.

DETAILED DESCRIPTION:
The investigators propose to use AZD1981 in subjects with chronic idiopathic urticaria (CIU) who are otherwise uncontrolled on first-line, oral antihistamine therapy. The skin lesion pathology in CIU shows a perivascular infiltrate of lymphocytes (both Th2 and Th1), eosinophils, and basophils, and closely resembles an allergen-induced late-phase reaction. Further, murine studies show that the chemoattractant receptor-homologous molecule expressed on Th2 (CRTh2) pathway is important in leukocyte recruitment following allergen challenge of the skin. Our proposed hypothesis is that AZD1981 in CIU will reduce CRTh2-expressing, leukocyte recruitment to the skin and reduce leukocyte activation through CRTh2, thus reducing the signs and symptoms in CIU refractory to control with antihistamines.

ELIGIBILITY:
Inclusion Criteria:

* Females must be surgically sterile or postmenopausal or using a highly effective form of birth control throughout the duration of the study
* Females must have a negative urine pregnancy test at screening
* Must meet the criteria for Chronic Idiopathic Urticaria (CIU) as defined by itching and hives for >3 days per week for over 6 weeks with no clear cause
* CIU symptoms must have started at least 6 months prior to starting the study
* Must have moderate to severe CIU, using a standardized survey, despite taking antihistamines

Exclusion Criteria

* Pregnant females or females who plan to become pregnant during the study
* Drug or alcohol abuse within the past 3 years
* Use of any investigational drug with 30 days of the start of the study
* Eczema or other skin conditions associated with itching (besides hives)
* Inability to comply with follow-up procedures
* Use of the following therapies in the past 30 days: hydroxychloroquine, sulfasalazine, dapsone, methotrexate, cyclophosphamide, Intravenous Immunoglobulin (IVIG), plasmapheresis, cyclosporine, oral or systemic steroids, or other monoclonal antibody therapies
* Use of doxepin within the past 2 weeks
* Use of either H2 antihistamines and leukotriene receptor antagonists within 7 days before starting the study (unless already on these medications for Gastroesophageal Reflux Disease (GERD), asthma or allergic rhinitis)
* Inability to take diphenhydramine (Benadryl)
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks or interfere with ability to comply with study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarbjit S Saini, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study involved a 1-week screening period and a 2-week single-blind placebo run-in before randomization to active or placebo treatment. 10/38 enrolled subjects were excluded based on low disease activity (n=5), inability to remain solely on daily H1 antihistamine (n=4), and noncompliance (n=1).
Groups:
- AZD1981: AZD1981 for oral administration will be available in tablet form. AZD1981 tablets will be provided in 10 mg strengths.
  The drug will be self-administered by the subject. Subjects will take 4 tablets in the morning, 4 tablets in the afternoon, and 4 tablets in the evening.
  The tablets should be swallowed whole with a glass of water.
  AZD1981: AZD1981 is an oral, potent, selective, reversible antagonist of CRTh2 (Chemoattractant Receptor Homologous Molecule expressed on Th2 cells).
- Placebo: The placebo will be available in tablet form. The placebo contains the same ingredients as the AZD1981 with the exception of the active compound.
  The placebo will be self-administered by the subject. Subjects will take 4 tablets in the morning, 4 tablets in the afternoon, and 4 tablets in the evening.
  The tablets should be swallowed whole with a glass of water.
  Placebo: Sugar pill manufactured to mimic AZD1981 10 mg tablet
Period: Overall Study
Arm/Group | AZD1981 | Placebo
Started | 14 | 14
Completed | 14 | 12
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants were randomized to AZD1981 or placebo at the end of placebo-run in, not at baseline. Values below reflect randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1981 | Placebo | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] — Population: There was no significant difference in age between study groups.
  years | 41.85 [23 to 65] | 45.17 [23 to 64] | 43.38 [23 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 12 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 4 | 8
  White | 6 | 4 | 10
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: The Change in Diary-based Clinical Symptoms as Measured by the Urticaria Activity Score 7 (UAS7)
Description: The UAS score, which is the sum of pruritus and hives, will be used to calculate the UAS7. UAS is a validated measure of Chronic Spontaneous Urticaria (CSU) disease activity which scores the intensity of pruritus (0-3, with 0 = no itch and 3 is severe itch) and number of hives (0-3 0 means no hives and 3 means greater than 50 hives) with a maximum value of 6 for a given day. The UAS7 is the sum of the daily average UAS scores (average of a.m. and p.m.) for 7 days with a minimum score of 0 and a maximum value of 42. The UAS7 is a sum of the daily average (average of a.m. and p.m.) for 7 days. The baseline score was established during the second placebo therapy week and compared to the final week of the 4 week active treatment period.
Time Frame: 7 Days
Population: One placebo subject had diary data compromised by device malfunction so only full data for 11 subjects were analyzed
Measure: Mean (Standard Error); unit: UAS7 Scores
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 12 | 11
UAS7 Scores
  Baseline | 20.46 (3.655) | 24.59 (3.463)
  End of Treatment | 18.83 (3.779) | 18 (3.614)
  End of Washout | 15.79 (3.726) | 19 (3.465)

2. Secondary Outcome: The Number of Participants With Adverse Events
Description: The safety of AZD1981 will be assessed using the following outcome measures: incidence and severity of treatment-emergent adverse events and serious adverse events, clinical laboratory measures, and vital signs. In particular we will measure CBC's with differential at baseline and week 4 and liver function tests every 2 weeks based on past trial experience of dose-related toxicity.
Time Frame: 8 weeks
Measure: Number; unit: participants with adverse events
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 14 | 12
participants with adverse events | 9 | 8

3. Secondary Outcome: The Ability of AZD1981 to Inhibit Prostaglandin D2 (PGD2)-Induced Eosinophil Shape
Description: The measure of Eosinophil shape change was assessed by cell scatter characteristics using a flow cytometer. Cellular scatter was established with buffer and then several doses of PGD2 stimulation.
Time Frame: Baseline, End of treatment, end of washout
Population: Insufficient samples were obtained for one active and 2 placebo patients.
Measure: Mean (Standard Deviation); unit: Mean fluorescence units area under curve
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 13 | 10
Mean fluorescence units area under curve
  Baseline | 1521.317 (138.146) | 1472.867 (184.401)
  End of Treatment | 1435.540 (137.752) | 1456.602 (157.485)
  End of Washout | 1508.367 (116.085) | 1406.221 (108.539)

ADVERSE EVENTS:
Arm/Group | AZD1981 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 9/14 | 8/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD1981 (N=14) | Placebo (N=12)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Infection (Infections and infestations) | 5 (5) | 5 (5)
Sleep impairment (Psychiatric disorders) | 1 (1) | 1 (1)
Respiratory disorders (non-infectious) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 5 (5) | 2 (2)
Blood disorders (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Eye and vision disorders (Eye disorders) | 0 (0) | 1 (1)
Cardiovascular disorders (Cardiac disorders) | 1 (1) | 1 (1)
Renal disorders (Renal and urinary disorders) | 0 (0) | 0 (0)
Reproductive disorders (Reproductive system and breast disorders) | 0 (0) | 0 (0)
Skin or hair disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Immunologic disorders (Immune system disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Among the limitations of this study are the small number of subjects, short duration of therapy and washout periods, and the lack of skin tissue biopsies to correspond with peripheral blood leukocyte findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No